CLINICAL TRIAL: NCT02696590
Title: Isfahan University of Medical Sciences
Brief Title: High Dose Oral Versus Intramuscular Vitamin D3 Supplementation In Multiple Sclerosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leila Dehghani, assistant prof, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Isfahan MS Society
Record Dates: First submitted 2016-02-18; First posted 2016-03-02 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MS patients injectable Vitamin D3 (Experimental): MS patients who received injectable form of Vitamin D3, received 600.000 IU Intramuscular vitamin D3 injection, in two weeks; 300.000 IU at the study entry and 300.000 IU in second week
  Interventions: Dietary Supplement: Vitamin D3
- MS patients orally Vitamin D3 (Experimental): received the same total dose of 600 000 IU D3 in two weeks, in the form of twelve pearls, each containing 50 000 IU D3 as follows: the first pearl was delivered at study entry, followed by one pearl each day for another 11 Days.
  Interventions: Dietary Supplement: Vitamin D3
- Healthy groups Injectable Vitamin D3 (Active Comparator): who received injectable form of Vitamin D3, received 600.000 IU Intramuscular vitamin D3 injection, in two weeks; 300.000 IU at the study entry and 300.000 IU in second week
  Interventions: Dietary Supplement: Vitamin D3
- Healthy groups Vitamin D3 orally (Active Comparator): received the same total dose of 600 000 IU D3 in two weeks, in the form of twelve pearls, each containing 50 000 IU D3 as follows: the first pearl was delivered at study entry, followed by one pearl each day for another 11 Days.
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — two forms of vitamin D3 (Oral versus injection) were compared in MS and healthy groups.
  Other Names: cholecalciferol

SUMMARY:
This study aimed to evaluate oral and injectable routes in treatment of hypovitaminosis D in multiple sclerosis (MS) patients. The investigators aimed to assess the efficacy of each method, using the same Mega dose of 600 000 IU D3, in achieving normal serum 25(OH)D level, the durability of the response, the practicality and the possible toxicity.

DETAILED DESCRIPTION:
Ultraviolet sunlight is too low to produce adequate amounts of vitamin D3, and vitamin D insufficiency lasting 4 to 6 months of the year at latitudes of ≥42° is common in individuals with low vitamin D intake. Vitamin D has strong immunoregulatory effects, and vitamin D supplementation prevents experimental autoimmune encephalomyelitis (EAE), an autoimmune disease in animals that is used as a model of MS.

Recently, emerging data from epidemiologic studies suggest that vitamin D may play an important role in the progression of the development of MS. A longitudinal study in pediatric MS showed a 34% lower risk of relapse for every 10 ng/ml higher 25-hydroxyvitamin D level. A similar magnitude of reduced relapse risk was later reported in an adult MS cohort. Higher vitamin D levels have also been shown to be associated with less subsequent inflammatory MS activity on brain magnetic resonance imaging (MRI). Finally, studies have demonstrated that patients have lower vitamin D levels during MS relapses.

ELIGIBILITY:
Inclusion Criteria:

* with serum 25(OH)D3 concentration ≤ 20 ng/ml

Exclusion Criteria:

* hypercalcaemia, primary hyperparathyroidism, Paget disease, thyrotoxicosis, pregnancy, active malignancy, hypercalciuria, history of liver disease, renal insufficiency, clinically apparent malabsorption syndrome, using drugs containing vitamin D products, calcium, estrogen and drugs known to affect vitamin D metabolism (anticonvulsants, glucocorticoids) or receiving any form of supplements containing vitamin D during last 6 months.
* Participants with serum 25(OH)D concentration≥ 20 ng/ml

Ages: 23 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2015-07; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Serum concentration of 25(OH)D | Two Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Masoud Etemadifar, professor, Study Director — Isfahan MS Society, Isfahan University of Medical Sciences, Isfahan, Iran
Locations (1):
- Alzahra Hospital, Isfahan, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Undecided